CLINICAL TRIAL: NCT00583089
Title: Decompensation Detection Study
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: DECODE
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Algorithm Test Set
- 2: Algorithm Development Set

SUMMARY:
To gather data and analyze decompensation events.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with an approved Guidant CRT-D HF device programmed to CRT therapy in VDD or DDD mode.
* Patients prescribed to the LATITUDE(R) system configured for at least weekly device interrogations and symptoms reporting.
* Patients willing to use the LATITUDE(R) enabled weight scale.

Exclusion Criteria:

* Patients that require adaptive rate pacing (rate-responsive modes).
* Patients that have received routinely scheduled intravenous inotropic therapy as part of their drug regimen within the past 90 days.
* Both

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 699 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Data collection and analysis. | End of patient follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Ewald, M.D., Principal Investigator — Washington University School of Medicine; F. Roosevelt Gilliam, M.D., Principal Investigator — Cardiology Associates of Northeast Arkansas